CLINICAL TRIAL: NCT02363452
Title: A Pilot Clinical Trial of Reverse Transcriptase Inhibitors in Children With Aicardi-Goutières Syndrome (AGS)
Brief Title: Reverse Transcriptase Inhibitors in AGS
Acronym: RTIs in AGS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P140203
Record Dates: First submitted 2015-01-15; First posted 2015-02-16 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Aicardi-Goutières Syndrome (AGS)
Keywords: Aicardi-Goutières syndrome; Reverse transcriptase inhibitors; open single study; interferon signature
MeSH Terms: interventions — Lamivudine; abacavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AGS (Experimental): Reverse transcriptase inhibitors
  Interventions: Drug: Reverse transcriptase inhibitors: Zidovudine, Lamivudine, Abacavir

INTERVENTIONS:
Drug: Reverse transcriptase inhibitors: Zidovudine, Lamivudine, Abacavir — Oral Solution (syrup) or Tablets

SUMMARY:
The purpose of this study is to determine if treatment with reverse transcriptase inhibitors returns the interferon signature observed in patients with AGS to normal levels.

DETAILED DESCRIPTION:
AGS is a genetically heterogeneous disease resulting from mutations in any one of the genes encoding the 3-prime repair exonuclease TREX1 (AGS1), the three non-allelic components of the RNASEH2 endonuclease complex (AGS2, 3 and 4), the Sam domain and HD domain containing protein (SAMHD1; AGS5) which functions as a deoxynucleoside triphosphate triphosphohydrolase, the double stranded RNA editing enzyme ADAR1, or the cytosolic dsRNA sensor IFIH1. It is hypothesized that AGS1-6 are involved in limiting the accumulation of intracellular nucleic acid species, a failure of which process results in triggering of an innate immune response that is more normally induced by viral nucleic acids. That is, in the absence of AGS-related protein activity, endogenous nucleic acids accumulate and are sensed as viral or 'non-self', leading to the induction of an interferon (IFN) alpha mediated immune response and the production of antibodies against self nucleic acids. AGS is associated with increased levels of interferon alpha in the cerebrospinal fluid (CSF) and serum. Available data suggest that AGS might be treated with (particular) reverse transcriptase inhibitors (which compounds can potentially disrupt both exogenous retroviral and endogenous retroelement cycling). No systematic approach to treatment in AGS has been explored. The investigators hypothesis is that reverse transcriptase inhibitors will also inhibit the reverse transcription of endogenous retroelements which are deemed to be responsible for initiating the tissue damage seen in AGS. Consequently, for the purpose of the investigators pilot study, it would be ideal to assess the effects of therapy by monitoring a reactive biomarker.

This is a single centre, open, single arm, phase II study in children with AGS. This study design is justified because no data are available about antiretroviral drug efficacy in children with AGS. Moreover, this study is the first step before a phase III study of drug efficacy.

The investigators propose a pilot clinical trial of selected reverse transcriptase inhibitors in AGS patients, with the specific endpoint of assessing the effect of treatment on the disease-associated interferon signature. The investigators propose to evaluate the safety of combination therapy comprising the three nucleoside analog reverse-transcriptase inhibitors (NRTIs) zidovudine (AZT), lamivudine (3TC), abacavir (ABC) in patients with AGS over a 52 week period of treatment. The inclusion period is 12 months. Patients can not participate in a biomedical trial of another drug during the 18 month follow-up (12 months of treatment period plus 6 months post treatment period).

A total of six visits (including a final visit) are scheduled for this trial over a period of 18 months (M1, M3, M6, M9, M12, M18) for all patients.

Drugs will be dispensed for medication at home, at usual doses recommended in HIV infection. Subjects will be dosed according to French guidelines. Dosing will be reviewed at each study visit against current weight, and modified as necessary in accordance with French dosing guidelines.

ELIGIBILITY:
Inclusion Criteria:

* A molecular diagnosis of AGS i.e. biallelic or known dominant mutations, with pathogenicity assessed using our extensive mutation database / functional data, in any of TREX1, RNASEH2A, RNASEH2B, RNASEH2C and SAMHD1 genes
* A pre-defined interferon signature (consistently present, moderate or high, on at least three occasions, over a period of 6 months prior to enrolment in the study)
* Age ≥ 1 month and < 18 years (either sex)
* Patient beneficiary or affiliated to " health insurance"
* Written informed consent

Exclusion Criteria:

* Pre-existing disease, not due to AGS, which would preclude the use of zidovudine, Lamivudine and abacavir (as currently assessed in routine clinical HIV-related practice)
* HLA B57-01 positive result, which indicates a greater risk of abacavir hypersensitivity reaction
* Patients with abnormally low neutrophile counts (<0.75 x 109/l), or abnormally low haemoglobin levels (<7.5 g/dl or 4.65 mmol/l)(zidovudine contraindication)
* Positive serology for HIV, HBV
* Known history of cirrhosis and history of clinically relevant hepatitis within last 6 months
* Moderate to severe renal impairment
* Pregnancy, breastfeeding
* Patient participating to a biomedical research with drug

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Interferon signature | Before and after 12 months of treatment
  Interferon Score

SECONDARY OUTCOMES:
Interferon signature | Month 18
  Interferon Score
Adverse Events | Baseline until Month 18
Interferon Activity Level in cerebrospinal fluid (UI/L) | Within the 12 month on treatment
Interferon Activity Level in blood (UI/L) | Within the 12 month on treatment
Interferon Activity Level in blood (UI/L) | month 18
Interferon Protein in cerebrospinal fluid (Fg/mL) | within the 12 month on treatment
Interferon Protein in blood (FG/mL) | Within the 12 month on treatment
Interferon Protein in blood (Fg/mL) | Month 18
Neurological assessment | Baseline
  Scale for Evaluation of Movement Disorders Vineland Adaptive Behaviour Scales
Neurological assessment | Month 12
  Scale for Evaluation of Movement Disorders Vineland Adaptive Behaviour Scales
Neurological assessment | Month 18
  Scale for Evaluation of Movement Disorders Vineland Adaptive Behaviour Scales
Radiological assessment | Baseline
  MRI, CT Scan
Radiological assessment | Month 12
  MRI, CT Scan
dosages of abacavir | Month 1
  Blood sample
dosages of zidovudine | Month 1
  Blood sample
dosages of lamivudine | Month 1
  Blood sample
dosages of zidovudine | Month 3
  Blood sample
dosages of lamivudine | Month 3
  Blood sample
dosages of abacavir | Month 3
  Blood sample
dosages of abacavir | Month 6
  Blood sample
dosages of zidovudine | Month 6
  Blood sample
dosages of lamivudine | Month 6
  Blood sample
Number of chilblains lesions | baseline
Number of chilblains lesions | Month 1
Number of chilblains lesions | Month 3
Number of chilblains lesions | Month 6
Number of chilblains lesions | Month 9
Number of chilblains lesions | Month 12
Number of chilblains lesions | Month 18

CONTACTS AND LOCATIONS:
Overall Officials: Yanick CROW, MD, PhD, Study Chair — Hôpital Necker - Enfants Malades Public Hospitals of Paris; Stéphane BLANCHE, MD,PhD, Principal Investigator — Hôpital Necker - Enfants Malades Public Hospitals of Paris
Locations (1):
- Hôpital Necker - Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crow YJ, Vanderver A, Orcesi S, Kuijpers TW, Rice GI. Therapies in Aicardi-Goutieres syndrome. Clin Exp Immunol. 2014 Jan;175(1):1-8. doi: 10.1111/cei.12115. PMID 23607857
- [Background] Rice GI, Meyzer C, Bouazza N, Hully M, Boddaert N, Semeraro M, Zeef LAH, Rozenberg F, Bondet V, Duffy D, Llibre A, Baek J, Sambe MN, Henry E, Jolaine V, Barnerias C, Barth M, Belot A, Cances C, Debray FG, Doummar D, Fremond ML, Kitabayashi N, Lepelley A, Levrat V, Melki I, Meyer P, Nougues MC, Renaldo F, Rodero MP, Rodriguez D, Roubertie A, Seabra L, Uggenti C, Abdoul H, Treluyer JM, Desguerre I, Blanche S, Crow YJ. Reverse-Transcriptase Inhibitors in the Aicardi-Goutieres Syndrome. N Engl J Med. 2018 Dec 6;379(23):2275-7. doi: 10.1056/NEJMc1810983. No abstract available. PMID 30566312